CLINICAL TRIAL: NCT02932865
Title: Modern Analyses of the Semen in Evaluating Male Fertility and Treatment Options of Male Infertility
Acronym: SemiFluid
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Lund University Hospital (Other); University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: SemiFluid
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Infertility, Male
Keywords: azoospermia; male fertility; MD-TESE; miRNA; piRNA; male infertility
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen sample Serum sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MD-TESE (A): Azoospermic men, MD-TESE operation (standard treatment). Semen sample, serum sample and physical examination with testicular ultrasound.
- Subfertile men (B): Subfertile men receiving medication (standard treatment). Semen sample, serum sample and physical examination with testicular ultrasound.
- Control (C): Control group, men scheduled for semen analysis. Semen sample, serum sample and physical examination with testicular ultrasound.

SUMMARY:
Men are recruited to collect seminal plasma samples and serum samples from men with azoospermia, men receiving medical treatment of infertility and men attending semen analysis. MicroRNA (miRNA) and PiWi-interacting RNA (piRNA) are analyzed for all of the groups to find potential differences. Steroid hormones are analyzed by liquid chromatography-tandem mass spectrometry.

DETAILED DESCRIPTION:
Azoospermic men attending microdissection testicular sperm extraction (MD-TESE) are group A. Second group (B) is the men with poor semen quality, who are treated with aromatase inhibitor, antiestrogen or human choriogonadotropic hormone (HCG) to improve semen quality. Third group (C) consists of men submitting semen analysis. The intended number of participants is 60, 60 and 100 men, respectively.

Seminal plasma and serum samples are collected and miRNA and piRNA are analyzed. Steroid hormones are analyzed by liquid chromatography-tandem mass spectrometry. The participants are given a physical examination and testicular ultrasound. The primary aim of this study is to develop a tool to better estimate the sperm recovery rate (SRR) of azoospermic men scheduled for MD-TESE. Since no data have been published presenting miRNA and piRNA levels in men with normal semen, a secondary aim is to describe the levels of miRNA and piRNA in unselected men. Third part of this study aims to find if medical treatment improving semen parameters affects miRNA ja piRNA findings.

ELIGIBILITY:
Inclusion Criteria:

* Ability to produce semen sample

Exclusion Criteria:

* Cognitive impairment
* Inadequate language skills for informed consent

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men contacting the fertility clinic in Turku University Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
miRNA and piRNA according to sperm recovery in MD-TESE | Two years

SECONDARY OUTCOMES:
Assess miRNA and pRNA changes with hormonal treatment | two years

OTHER OUTCOMES:
Describe miRNA and piRNa levels in seminal plasma of unselected men | two years

CONTACTS AND LOCATIONS:
Overall Officials: Antti Perheentupa, MD,PhD, Study Director — University of Turku
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No